CLINICAL TRIAL: NCT04410861
Title: Comparison of Panmacular Versus Minimal Micropulse Laser Therapy in Central Serous Chorioretinopathy
Brief Title: Panmacular Versus Minimal Micropulse Laser Therapy in Central Serous Chorioretinopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Moorfields Eye Hospital Centre Abu Dhabi (Other)
Collaborators: University of Warmia and Mazury in Olsztyn (Other); University of Gdansk (Other); The Filatov Institute of Eye Diseases and Tissue Therapy (Other); Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Igor Kozak, Consultant Vitreoretinal Surgeon/Clinical Lead, Moorfields Eye Hospital Centre Abu Dhabi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MoorfieldsEyeAbuDhabi
Record Dates: First submitted 2020-05-27; First posted 2020-06-01 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Central Serous Chorioretinopathy
MeSH Terms: conditions — Central Serous Chorioretinopathy

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Minimal Micropulse Arm (Active Comparator): Wavelength 810 577 Power 0.75 W 0.15 W DC 5% 5% Spot size 125um 100um Duration 0.3 sec 0.3 sec Number of spots 100-120 100-120
  .
  Interventions: Procedure: Micropulse laser photostimulation
- Panmacular Micropulse Arm (Experimental): Wavelength 810 577 Power 1.7 W 0.425 W DC 5% 5% Spot size 500um 500um Duration 0.3 sec 0.3 sec Number of spots 400-450 400-450
  Interventions: Procedure: Micropulse laser photostimulation

INTERVENTIONS:
Procedure: Micropulse laser photostimulation — In this treatment invisible, non-damaging laser shots are delivered to the affected area which are believed to lead to absorption of accumulated retinal fluid. Contact lens will be used along with topical anesthesia.Following the procedure eye will be washed with balanced salt solution.

SUMMARY:
Central serous retinopathy is a disease of poorly understood etiology characterized by accumulation of subretinal fluid and leading to significant decrease in vision. Micropulse laser therapy has been successfully used in the treatment of CSR of both acute and chronic types (1). In this treatment invisible, non-damaging laser shots are delivered to the affected area which are believed to lead to absorption of accumulated fluid. The mechanism of fluid resorption is unclear. There are several treatment protocols in place (2, 3). Most commonly reported are minimal protocol and so-called panmacular protocol. However, there is no comparative study between them assessing their clinical efficacy.

The purpose of this trial is to compare treatment efficacy in central serous chorioretinopathy (CSR) using two laser parameter settings. Those will include minimal and panmacular protocols. Two wavelengths will be used 577nm and 810 nm for which the rest of the parameters will be defined in order to produce sublethal photostimulation. Structural and functional outcomes will be compared before and after treatment as well as measures such as number of repeat treatments or need for rescue treatment. We aim to show which of the laser arms will lead to better clinical outcomes.

DETAILED DESCRIPTION:
Study Design:

This is a comparative, prospective, interventional, multicenter, randomized study of micropulse laser treatment of central serous chorioretinopathy with 2 treatment arms:

1. < 6 months. Treatment: Minimal vs. Panmacular (randomized)
2. > 6 months. Treatment: Panmacular only

Treatment arms - description of laser settings:

For "Minimal / PLACE" treatment (Mainster contact lens with magnification of 1.05x):

Wavelength 810nm or 577nm, Power 0.75 Watt for 810 nm or 0.15 Watt for 577 nm, Duty Cycle 5% for both wavelenths, Spot size 125um for 810 nm and 100um for 577 nm, Duration 0.3 sec 0.3 sec for both wavelenths, Number of spots 100-120 for both wavelenths

For "Panmacular" treatment (Mainster lens mag 1.05x):

Wavelength 810nm or 577nm, Power 1.70 Watt for 810 nm or 0.425 Watt for 577 nm, Duty Cycle 5% for both wavelenths, Spot size 50um for both wavelengths, Duration 0.3 sec 0.3 sec for both wavelenths, Number of spots 400-450 for both wavelenths

All treatments will be performed following informed consent and under topical anesthesia using eyedrops 3x before procedure in the treatment eye(s). Follow-up will be every 6 weeks with final one in 6 months. Each follow-up visit will include visual acuity measurement, intraocular pressure, slit-lamp examination, VF and OCT examinations.

Primary Endpoints:

1. Visual Acuity as measured by ETRDS chart (number of letters before and after treatment
2. Complete subretinal fluid resolution as assessed by OCT examination (microns of central retinal thickness before and after treatment; presence/absence of subretinal fluid)

Secondary Endpoints:

1. Visual Field - Humphrey 10-2 protocol (dB value before and after treatment)
2. Number of treatments required for vision/structure improvement (number of laser sessions)
3. Rescue rate - number of eyes requiring intravitreal injection of anti-angiogenic agents or oral eplerenone

Risks: Non-response to therapy in which case alternative rescue treatments (intravitreal injection or oral eplerenone) will be offered to patient.

Benefits: Patient participating in the study will receive standard of care. Participation will be entirely voluntary and in case of withdrawing from the study patient will be receiving alternative approved methods of treatment.

ELIGIBILITY:
Inclusion Criteria:

* CSR diagnosed < 6 months ago Willingness to undergo micropulse laser treatment and keep follow-up visits

Exclusion Criteria:

* High myopia Other significant macular disease, other treatment for CSR Pregnancy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in Best-Corrected Visual Acuity (BCVA) | 6 months
  BCVA will be measured using ETDRS charts and number of letters will be compared before treatment and during follow-up and at the last visit.
Resolution of Subretinal Fluid | 6 months
  This outcome will be assessed by optical coherence tomography (OCT). Microns of central retinal thickness will be compared before treatment and during follow-up and at the last visit. The presence/absence of subretinal fluid will be recorded.

SECONDARY OUTCOMES:
Visual Field Examination | 6 months
  This will be assessed by Humphry VF analyzer - 10-2 protocol and dB values will be compared before treatment, during follow-up and at the last visit.
Need for Re-treatment | 6 months
  The number of eyes which have nor responded to micropulse treatment and required rescue treatment either intravitreal injection of anti-angiogenic agent or oral eplerenone will be recorded and compared between laser groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Moorfields Eye Hospital Centre, Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No
Due to patient confidentiality we do not plan to share individual patient data

REFERENCES:
- [Background] Chhablani J, Roh YJ, Jobling AI, Fletcher EL, Lek JJ, Bansal P, Guymer R, Luttrull JK. Restorative retinal laser therapy: Present state and future directions. Surv Ophthalmol. 2018 May-Jun;63(3):307-328. doi: 10.1016/j.survophthal.2017.09.008. Epub 2017 Oct 5. PMID 28987614
- [Background] Kozak I, Luttrull JK. Modern retinal laser therapy. Saudi J Ophthalmol. 2015 Apr-Jun;29(2):137-46. doi: 10.1016/j.sjopt.2014.09.001. Epub 2014 Sep 28. PMID 25892934
- [Result] Wood EH, Karth PA, Sanislo SR, Moshfeghi DM, Palanker DV. NONDAMAGING RETINAL LASER THERAPY FOR TREATMENT OF CENTRAL SEROUS CHORIORETINOPATHY: What is the Evidence? Retina. 2017 Jun;37(6):1021-1033. doi: 10.1097/IAE.0000000000001386. PMID 27841848